CLINICAL TRIAL: NCT05627804
Title: Effects of Normobaric Hypoxia and Different Exercise Modes on Blood Glucose Regulation in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Collaborators: National Sports Institute of Malaysia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ISNRP-003-2020
Record Dates: First submitted 2022-11-13; First posted 2022-11-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Overweight; Healthy; Physical Inactivity
MeSH Terms: conditions — Overweight; Sedentary Behavior | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate hypoxia (Experimental): The participant will perform different exercise modes under moderate hypoxia (fraction oxygen: 16.5%). Blood samples immediately after exercise oral glucose tolerance test will be collected.
  Interventions: Other: Low-moderate intensity exercise; Other: Sprint interval training; Other: Functional exercise
- Control normoxia (Other): The participant will not perform any exercise under normoxia and moderate hypoxia. Blood samples of oral glucose tolerance test will be collected.
  Interventions: Other: Control

INTERVENTIONS:
Other: Low-moderate intensity exercise — The participants will perform low-intensity cycling exercise at 90% lactate threshold under moderate hypoxia
  Arms: Moderate hypoxia
Other: Sprint interval training — The participants will perform sprint interval cycling exercise at a load of 7.5% bodyweight under moderate hypoxia.
  Arms: Moderate hypoxia
Other: Functional exercise — The participants will perform bodyweight exercises under moderate hypoxia.
  Arms: Moderate hypoxia
Other: Control — No exercise will be performed.
  Arms: Control normoxia

SUMMARY:
Obesity is a major global health issue and a primary risk factor for metabolic-related disorders. While physical inactivity is one of the main contributors to obesity, it is a modifiable risk factor with exercise training as an established, non-pharmacological treatment to prevent the onset of metabolic-related disorders, including obesity. Exposure to low-oxygen availability (hypoxia) via normobaric hypoxia (simulated altitude via reduced inspired oxygen fraction), termed hypoxic conditioning, in combination with exercise has been increasingly shown in the last decade to enhance blood glucose regulation and decrease body mass index, providing a feasible strategy to treat obesity.

However, findings from studies investigating the potential for hypoxia to augment the exercise training response and subsequent metabolic health are equivocal. Notably, there is a lack of information regarding the optimal combination of exercise variables and hypoxic severity to enable an individualized and safe practice of exercising in a hypoxic environment.

In the present randomized, single-blind, cross-over study, the investigators will investigate the effects of single-bout of different exercise modes under moderate hypoxia (FiO2, 16.5%).

The investigators hypothesize that all exercises combined with hypoxia improve glucose homeostasis in overweight individuals.

DETAILED DESCRIPTION:
In the present randomized, single-blind, cross-over study, participants will be exposed to moderate hypoxia (oxygen level 16.5%) during three different exercises (low-intensity cycling, sprint interval and functional exercises). Participants will be randomly assigned to each exercise condition (computer-generated randomization plan), separated by a washout period (5-7 days). To accomplish this, participants will exercise in an environmental chamber in which oxygen concentration of the ambient air and, as such, oxygen levels can be closely controlled and monitored.

Participants are required to attend the laboratory 8 times. These visits are including pre-exercise screening, baseline blood sampling, body composition screening and exercise in altitude conditions.

ELIGIBILITY:
Inclusion Criteria:

* BMI is between 25-29 kg/m²
* Physical inactive (physical activity <150 min/week)
* No known heart or metabolic diseases (such as Type 2 diabetes)
* Not currently taking any prescribed medication
* No reported musculoskeletal injuries recently
* Not exposed to hypoxia >1000 m prior to the study

Exclusion Criteria:

* Impaired glucose tolerance (2 hour glucose: >7.8 - 11.1 mmol/L)
* Type 2 diabetes mellitus
* Obstructive sleep apnea
* Chronic obstructive pulmonary disease

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Oral glucose tolerance test (glucose) | Change of fasting and postprandial plasma glucose concentrations compared to different exercise mode at immediately after exercise
  Change of plasma glucose concentration immediately post-exercise under different exercise modes
Oral glucose tolerance test (insulin) | Change of fasting and postprandial plasma insulin concentrations compared to different exercise mode at immediately after exercise
  Change of plasma insulin concentration immediately post-exercise under different exercise modes

CONTACTS AND LOCATIONS:
Locations (1):
- National Sports Institute of Malaysia, Kuala Lumpur, Malaysia